CLINICAL TRIAL: NCT00625638
Title: Symptom Assessment in Advanced Cancer Patients Using an Interactive Voice Response (IVR) System
Brief Title: Interactive Voice Response System in Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0591; NCI-2012-01747 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Caregiver; Interactive Voice Response; Symptom Control; IVR System; Questionnaire
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Only (Experimental): Participants will return with the caregiver on day 15 to complete a questionnaire lasting 30 minutes.
  Interventions: Other: Standard Care
- Standard Care + IVR System (Experimental): Standard Care + Interactive Voice Response (IVR) System Participants will return with the caregiver on day 15 to complete a questionnaire lasting 30 minutes. Phone calls made once daily, each taking about 3-5 minutes to complete.
  Interventions: Behavioral: Interactive Voice Response System; Other: Standard Care

INTERVENTIONS:
Behavioral: Interactive Voice Response System — Phone calls made once daily, each taking about 3-5 minutes to complete.
  Arms: Standard Care + IVR System
Other: Standard Care — Participants will return with the caregiver on day 15 to complete a questionnaire lasting 30 minutes.

SUMMARY:
The goal of this research study is to learn if using an Interactive Voice Response (IVR) system can bring about better and more timely symptom control for patients with advanced cancer.

Primary Objectives:

* To determine whether the Interactive Voice Response (IVR) system, supplemented by Nursing Telephone Intervention (NTI), results in better symptom management and quality of life than standard care for individuals with advanced cancer as evidenced by reduced scores on symptom measures.
* To determine whether the IVR system, supplemented by NTI, results in reduced caregiver burden, increased caregiver satisfaction with care, and improved coping strategies.
* To determine the feasibility of using an IVR system, supplemented by NTI, for symptom assessment in individuals with advanced cancer and their caregivers by conducting a process evaluation of the system. Variables to be evaluated include rates of participant recruitment and retention, frequency of use of the system, acceptability of the system to participants, and barriers to participation. Researchers' goal is to identify and improve aspects that affect external validity (recruitment rate, cohort maintenance), internal validity (implementation, contamination), participant acceptability and satisfaction, and reaction to study procedures. The findings from this evaluation will also allow researchers to evaluate delivery of interventions in future studies.

DETAILED DESCRIPTION:
If you and your caregiver agree to take part in this study, you will be randomly assigned (as in the toss of the coin) to be in 1 of 2 groups. Group A will receive standard of care provided at the palliative center at M. D. Anderson, but will not receive any phone calls from the Interactive Voice Response (IVR) system. Group B will receive phone calls by the Interactive Voice Response (IVR) system on Monday, Wednesday, and Friday for 15 days.

Once you sign this consent form, you will answer questions about your diagnosis, the medication that you take, and the symptoms that you are having (for example, pain, fatigue, anxiety, depression, and overall feeling of well-being). You will either be asked these questions verbally or you will complete a written questionnaire. This should take about 30 minutes to complete.

If you and your caregiver are assigned to Group A, you will continue with the standard of care provided at the palliative center at M. D. Anderson. On Day 15, both you and your caregiver will be seen in the outpatient clinic by the research nurse, and complete the same questionnaire you had at the beginning of the study, either verbally or written. This should take about 30 minutes to complete.

If you and your caregiver are assigned to Group B, a research nurse will train you and your caregiver to operate the IVR system. The IVR call will be made to the preferred telephone number(s) provided by you and your caregiver. The telephone calls will be made 1 time a day at times chosen by you and your caregiver. You will both be given a 3-digit code number to enter as a way of confirming who you are.

Once you have entered the requested numbers, the IVR system will ask you to answer questions about pain, fatigue, anxiety, depression, and your overall feeling of well-being. These phone calls should take about 3-5 minutes to complete. You should complete the phone calls separately and should not attempt to influence each others answers.

A research nurse will review the answer in the IVR system. If you haven't responded to the IVR questions in 3 days, if you answer that you would like to be contacted by a nurse, or if a symptom has reached a concerning level, you and your caregiver will receive a phone call from the nurse. The nurse may ask about symptoms, medications being taken, concerns or doubts about the medication, and if you have any concerns about your physical or emotional well being. You will be reminded of the different telephone numbers you can use to receive assistance 24 hours a day. During the phone call, you will also be asked if you would like the nurse to contact your caregiver for information and support. If you agree, the nurse will contact your caregiver.

On Day 8, both you and your caregiver will be contacted either in person or by phone by the research nurse and will complete the same questionnaire you had at the beginning of the study. On Day 15, both you and your caregiver will be seen in the outpatient clinic by the research nurse and will complete this same questionnaire again, either verbally or written. This should take about 30 minutes to complete each time.

Your participation on this study will end on Day 15.

This is an investigational study. Up to 68 patient-caregiver groups (or a total of 136 participants) will take part in this study. All the participants will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with advanced cancer (incurable disease) who are seen in the Supportive Care Center at M.D. Anderson Cancer Center.
2. Individuals with advanced cancer who have a pain score of 4 or higher on the average pain scale item of the Brief Pain Inventory for at least 2 weeks
3. Individuals with advanced cancer who have a score of 4 or higher on pain and at least one other symptom on the ESAS (fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep).
4. Individuals with advanced cancer who are able to identify a primary caregiver who also agrees to participate in the study
5. Individuals with advanced cancer who have no clinical evidence of cognitive failure in the opinion of the referring MD.
6. Individuals with advanced cancer and caregivers who are at least 18 years of age
7. Individuals with advanced cancer and caregivers who have access and utilize a touch-tone telephone
8. Individuals with advanced cancer and caregivers who are willing to engage in a telephone follow-up with the IVR system and nurses every Monday, Wednesday and Friday.
9. Individuals with advanced cancer and caregivers who are willing to follow-up by phone or in person on day 8 (+/- 3 days) and return for a follow-up visit on day 15 (+/-5 days)
10. Individuals with advanced cancer and caregivers who are willing and able to provide written informed consent
11. Must be English speaking [The IVR only available in English]
12. Caregiver must be a partner, parent, sibling, or child of the individual with advanced cancer.
13. Caregiver must reside with the individual with advanced cancer and be responsible for most of the individual with advanced cancer's care
14. Individuals with advanced cancer and caregivers must be able to understand the instructions for the study

Exclusion Criteria:

1. Individuals with advanced cancer or caregivers who cannot complete the baseline assessment forms
2. Individuals with advanced cancer or caregivers who cannot understand the requirements for participation in the study
3. Individuals with advanced cancer or caregivers who have hearing or visual impairments severe enough to prevent use of the IVR or Nursing Telephone Intervention (NTI)
4. Individuals with advanced cancer or caregivers who cannot understand and speak English (The IVR is only available in English)
5. Individuals with advanced cancer with caregivers who refuse to participate in the study
6. If individuals with advanced cancer are found to screen positive for severe mood disorders according to the HADS questionnaire for anxiety and/or depression, [ >/= to 20], they will be immediately referred to their primary palliative care physician for initial assessment and management including potentially a referral to psychiatry. Participants that are referred for psychiatric evaluation will be excluded from the study.
7. Caregivers who are suspected to have severe mood disorders will be instructed to contact their personal physician for assessment and management including potentially a referral to psychiatry. Those that are referred for psychiatric evaluation will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2008-01-28 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Determine if follow up by an IVR system results in better symptom management and improved quality of life for participants than standard care. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org